CLINICAL TRIAL: NCT06943196
Title: Effects of Structured Physical Activity Breaks and Free Play in Classroom on Gross Motor Skills, Endurance, and Behavior in Children With Mild Intellectual Disability
Brief Title: Effects of Structured Physical Activity Breaks and Free Play in Children With Mild Intellectual Disability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR/AHS/24/0739
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Intellectual Disability, Mild
Keywords: Endurance; Behavior; Neurodevelopmental disorder
MeSH Terms: conditions — Intellectual Disability; Lymphoma, Follicular; Behavior; Neurodevelopmental Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Structured physical activity break (Experimental): The structured physical activity breaks in classroom will include 5-30 minutes physical activities sequenced as: Week 1,4,7: 5-mintue stretch break, 5-minute marching in place, 30-sec jumping an invisible rope, 30-sec Flap arms like a bird, 5-minute mirror each other's actions and guess, 5-minute hop on one foot/ jump on both feet, draw on board, guess the color, make a circle and play a game of throw a ball in class. Week 2,5,8: 5-minute stretch break, 2-3 laps throughout the classroom, jumping in and out a circle on command, rock-paper-scissors-jump, paint or sketch on book, guess the animal, up-down-stop-go opposites, make a circle and play a game of throw a ball and clap in class.
  Week 3,6: 5-minute stretch break, 30-sec balance on one foot, 30-sec hopping, 5-jumping jacks, 5-claps turn around and guess the shape, play a game on board or notebook, make a circle and play a game of throw a ball and jump in class.
  Interventions: Other: Structured physical activity break
- Free play (No Intervention): Free play in classroom will be the activity stations available in the institute.
  Classroom will be divided into various zones, offering the widest selection of areas for the children to explore. Each zone will have age-appropriate play stations designed to engage the children in diverse activities. In addition to all of the locations, a reserve spots in the classroom will be made so that the students can show their work. This comprises the artwork and crafts that kids will have created in the free play classroom. Free Play is children's self-organized activity. Therapist will observe children in a creative, stimulating play environment and participation in the play.

INTERVENTIONS:
Other: Structured physical activity break — The structured physical activity breaks in classroom will include 5-30 minutes physical activities sequenced as: Week 1,4,7: 5-mintue stretch break, 5-minute marching in place, 30-sec jumping an invisible rope, 30-sec Flap arms like a bird, 5-minute mirror each other's actions and guess, 5-minute hop on one foot/ jump on both feet, draw on board, guess the color, make a circle and play a game of throw a ball in class. Week 2,5,8: 5-minute stretch break, 2-3 laps throughout the classroom, jumping in and out a circle on command, rock-paper-scissors-jump, paint or sketch on book, guess the animal, up-down-stop-go opposites, make a circle and play a game of throw a ball and clap in class.
  Week 3,6: 5-minute stretch break, 30-sec balance on one foot, 30-sec hopping, 5-jumping jacks, 5-claps turn around and guess the shape, play a game on board or notebook, make a circle and play a game of throw a ball and jump in class.
  Arms: Structured physical activity break

SUMMARY:
Children with mild intellectual disability (MID) typically exhibit delays in both intellectual and adaptive functioning, with the onset occurring during the developmental period.

These children often learn new information and skills at a slower pace compared to their peers and frequently struggle academically. Structured physical activity breaks (SPAB) in the classroom are short, planned periods of physical exercise integrated into the school day to enhance children's physical fitness and behavioral outcomes. Free play (FP) in which children may choose and engage in activities at their own pace, establishing creativity, social engagement, and self-regulation. Study includes 22 participants and divided into 2 groups, one group receiving (SPAB) and the other group participating in free play (FP). The physical activity breaks, lasting between 5 to 30 minutes. SPAB group will engage in a sequence of activities. These activities will start with a 5-minute stretch, followed by 5 minutes of marching in place, 30 seconds of jumping an invisible rope, 30 seconds of flapping arms like a bird, 5 minutes of mirroring each other's actions and guessing, 5 minutes of hopping on one foot or jumping on both feet, drawing on the board, guessing the color, and making a circle to play a game in class. In comparison, the FP group will have access to various activity stations within the classroom, allowing children to choose their activities within a 30-minute time frame. The intervention will be implemented 5-days a week for a total of 8-weeks. Gross Motor Development-2 (TGMD-2) use for assessing gross motor skills, the 6-minute walk test use for measuring functional capacity of endurance, and the Strengths and Difficulties Questionnaire (SDQ) use for evaluating behavior. Data analysis will be conducted using SPSS version 27.

DETAILED DESCRIPTION:
Children with mild intellectual disability (MID) typically exhibit delays in both intellectual and adaptive functioning, with the onset occurring during the developmental period. These children often learn new information and skills at a slower pace compared to their peers and frequently struggle academically. Structured physical activity breaks (SPAB) in the classroom are short, planned periods of physical exercise integrated into the school day to enhance children's physical fitness and behavioral outcomes. Free play (FP) in which children may choose and engage in activities at their own pace, establishing creativity, social engagement, and self-regulation. Gross motor skills, which include activities such as running, jumping, and balancing, are crucial for the overall physical development of children. Endurance, the ability to sustain physical activity over time often underdeveloped in children with MID. Behavioral outcomes, including social interaction, attention, and self-control, are also influenced by physical activity. This study aims to investigate the comparative effects of implementing SPAB as part of a comprehensive school physical activity program and FP on children with mild intellectual disabilities. Study includes 22 participants and divided into 2 groups, one group receiving (SPAB) and the other group participating in free play (FP). The physical activity breaks, lasting between 5 to 30 minutes. SPAB group will engage in a sequence of activities. These activities will start with a 5-minute stretch, followed by 5 minutes of marching in place, 30 seconds of jumping an invisible rope, 30 seconds of flapping arms like a bird, 5 minutes of mirroring each other's actions and guessing, 5 minutes of hopping on one foot or jumping on both feet, drawing on the board, guessing the color, and making a circle to play a game in class. In comparison, the FP group will have access to various activity stations within the classroom, allowing children to choose their activities within a 30-minute time frame. The intervention will be implemented 5-days a week for a total of 8-weeks. Gross Motor Development-2 (TGMD-2) use for assessing gross motor skills, the 6-minute walk test use for measuring functional capacity of endurance, and the Strengths and Difficulties Questionnaire (SDQ) use for evaluating behavior. Data analysis will be conducted using SPSS version 27.

ELIGIBILITY:
Inclusion Criteria:

* Mild Intellectual Disability i-e mild deficit in intellectual and adaptive functions, having onset in developmental period (24) approximate IQ range of 50 to 69 (25).
* ADLs are preserved and complex functions minimally impaired (26).
* Attendance of a special educational center;
* A medically cleared status from any physical ailment for participation in the baseline examinations.
* Children are able/ allowed to interact with the environment and use of resources during free play in school/institute

Exclusion Criteria:

* Children with chronic medical conditions/ physical disabilities/balance issues/injuries that prevent participation in physical activity
* Lack of informed consent from parents' and/or legal guardians' for their children's participation;
* Coexisting conditions: autism, Down syndrome, cerebral palsy (CP), any muscular dystrophy, or neurological disorders such as epilepsy or brain damage;
* Children with severe motor disability Comorbidities like oncological, rheumatic, orthopedic or cardiac diseases

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2025-04-17 (Actual); Primary Completion 2025-09-17 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
TGMD-2 for Gross Motor Skills | 8-weeks.
  "TGMD-2" is a tool for gross motor skills evaluation (30) and physical activity (31) in school age children. It comprises of two subtest categories locomotion to measure ability of child to move from one place to another, object control subtest measure the ability of child to perform object manipulation and visual-motor skills. The locomotor subtest has a maximum score of 48 (6 skills × 4 criteria x 2 trials), as does the object control subtest.
  The overall TGMD score is the sum of the two subgroups and it ranges from 0 to 96, with higher scores signifying better performance. To calculate the child's percentile rank and standard score, compare the total scores to the normative data in the TGMD-2 manual.
6MWT for endurance | 8-weeks
  "6-minute walk test" is a tool for measuring functional endurance and physical fitness. Six minute walk test (6MWT) is a field exercise test widely used in clinical practice both in adults and in pediatric patients. Anthropometric characteristics are measured before the test and, peripheral oxygen saturation (SpO2), heart and respiratory rate are measured before and after a 6-minute walk test
Strengths and Difficulties Questionnaire for behavior | 8-weeks
  "Strengths and Difficulties" Parent and Teacher reported questionnaire for children aged 04-17 years is a behavioral measuring tool. The SDQ includes 25 items that examine a range of 'strengths and difficulties' as behavioral indicators of probable mental health disorders. The items contribute to 5 subscales, each with 5 items and a minimum score ranging from 0 (lowest score) to 10 (highest score): conduct difficulties, hyperactivity/inattention, emotional signs, problems with peers, and social conduct. The sum of the first 4 subscales, a total difficulty score that ranges from 0 to 40 (40).

CONTACTS AND LOCATIONS:
Overall Officials: Maria Amjad, MSPT(Peads), Principal Investigator — Riphah International University
Locations (1):
- PSRD, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No